CLINICAL TRIAL: NCT04645420
Title: Molecular Effects of Apremilast in the Synovium of Psoriatic Arthritis Patients (MEAS Study)
Brief Title: Molecular Effects of Apremilast in the Synovium of Psoriatic Arthritis Patients
Acronym: MEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P1200_46; AP-CL-PSA-PI-13146 (Other Grant/Funding Number: AMGEN); 2019-003887-39 (EudraCT Number); 2020/24AOU/424 (Other: Ethic committee - Institutional Review Board)
Record Dates: First submitted 2020-10-30; First posted 2020-11-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psoriatic Arthritis
Keywords: Biologics; Apremilast; Synovium; Genomics; Psoriatic disease
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apremilast (Experimental): 15 PsA patients with active disease and naïve to conventional synthetic and biologic disease modifying anti-rheumatic drugs.
  Treatment with apremilast orally in the whole group (n = 15). Escalating dose the first Week (10 mg once day1, 10 mg bid day2, 10 mg-20 mg day3, 20 mg bid day4, 20 mg-30 mg day5, 30 mg bid on day6), and 30 mg bid from day7 until week24.
  Interventions: Procedure: Global gene expression profiles obtained from synovial biopsies.

INTERVENTIONS:
Procedure: Global gene expression profiles obtained from synovial biopsies. — Global gene expression profiles obtained from synovial biopsies before and after 24 weeks of treatment with the drug in each patient.
  Other Names: No other intervention

SUMMARY:
This study assess the genomics profiles in synovial biopsies obtained prior to, and 24 weeks after an immunomodulator agent (Apremilast) in patients with active psoriatic arthritis who are naive to treatment with a conventional synthetic DMARDs (such as methotrexate).

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1 BACKGROUND Psoriasis and Psoriatic Arthritis Psoriasis is a chronic relapsing immunologically mediated skin disease manifesting as red scaly plaques, which affects about 1-3% of the population.(ref.1-3). Ten to 20% of the people with psoriasis may develop an arthropathy, which affects small or large joints in a symmetrical or asymmetrical fashion(ref.4). Psoriatic arthritis (PsA) is the second most common inflammatory arthritis after rheumatoid arthritis, accounting for 10% to 15% of the patients attending early arthritis clinics(ref.5).

   PsA is a heterogeneous disease affecting 0.3 to 1% of the population(ref.6) and recent evidence showed significant disability if this condition is not adequately treated. About 15-35% had marked limitations of their functional capacity. Moreover patients with PsA have an increased mortality risk compared to the general population. A 59 and 65%-increased death rate was seen among respectively male and female PsA patients(ref.7).

   Different systemic treatments such as sulfasalazine, leflunomide, methotrexate, and biologics are widely used to treat PsA (ref.8) but not all patients respond to or tolerate these treatments. In addition, not all manifestations of PsA (like joints, dactylitis, scalp, enthesitis, or nails) may respond equally well.

   Apremilast Mechanism of action and indications Otezla (apremilast) is an innovative oral small-molecule inhibitor of phosphodiesterase (PDE) 4 that works intracellularly to modulate a network of pro- and anti-inflammatory mediators (ref.9,10). PDE4 is a cyclic adenosine monophosphate (cAMP)-specific PDE and is the dominant PDE in inflammatory cells. Inhibition of PDE4 elevates intracellular cAMP levels, which in turn down-regulates the inflammatory response by modulating the expression of tumour necrosis factor alpha (TNF-α), interleukin (IL)-23, IL-17, and other pro-inflammatory cytokines. Elevation of cAMP also increases anti-inflammatory cytokines. These pro- and anti-inflammatory mediators have been implicated in psoriasis and PsA. The pro-inflammatory mediators that are upregulated in PsA include the cytokines TNF-α, IL-1, IL-6, and IL-8, and the chemokines monocyte chemotactic protein-1 and macrophage inflammatory protein-1 beta (ref.9,11-13,17).

   Based on these effects, apremilast has been developed for use in the treatment of various immune-mediated inflammatory conditions such as psoriasis and PsA and it is under investigation in Behçet disease. A total of 4,089 patients have been exposed to apremilast across multiple indications, including 1,945 patients in the PsA Phase 3 clinical program (PALACE program)(Ref.14) and 1,184 patients in the psoriasis Phase III clinical program (ESTEEM program)(Ref.15,16).

   Otezla was approved in Europe in January 2015 for the treatment of active PsA, alone or in combination with disease modifying antirheumatic drugs (DMARDs), in adult patients who have had an inadequate response or who have been intolerant to a prior DMARD therapy (Ref.17). In the same time, Otezla was approved for the treatment of moderate to severe chronic plaque psoriasis in adult patients (≥18 years) who failed to respond to, or who have a contraindication for, or are intolerant to other systemic therapy including cyclosporine, methotrexate or psoralen and ultraviolet-A light. The recommended dose is 30 mg twice daily following an initial up-titration phase of 5 days. Otezla is administered orally, without regard to meals.

   Summary of efficacy and safety data Efficacy and safety of apremilast in the treatment of patients with active PsA who were inadequately controlled by DMARDs and/or biologics have been demonstrated in 3 multi-centre, randomised, double-blind, placebo-controlled trials (PALACE 1, 2, and 3) (Ref. 6,13,14,17). Results from these trials showed that apremilast treatment with or without concomitant DMARDs, compared with placebo with or without concomitant DMARDs, resulted in greater improvement in the signs and symptoms of PsA and more specifically in dactylitis and enthesitis in patients with these pre-existing symptoms, and these improvements were sustained. In clinical trials with apremilast, the majority of the most common adverse reactions occurred within the first 2 weeks of treatment and tended to resolve over time with continued dosing. The most frequently observed adverse reactions leading to discontinuation after 16 weeks of treatment with Otezla 30 mg twice daily were nausea, diarrhoea, and headache. Recently, reports of suicidal ideation and depression have been published, prompting more rigorous evaluation of the risk: benefit ratio and monitoring (Ref.18).

   1.2 STUDY RATIONALE Psoriatic arthritis is a chronic inflammatory disease, leading to impaired function and a reduced quality of life. Fortunately, improved knowledge about disease mechanisms has catalyzed rapid development of effective targeted therapies for this disease (Ref.19).

   Our laboratory has gained international recognition in the evaluation of transcriptomic patterns of synovial biopsies from patients with arthritis. Our work not only led to the identification of disease-specific molecular patterns in synovial tissue from patients with early rheumatoid arthritis (RA) (Ref.20,21), and the development of a diagnostic kit (Rheumakit®), but also to the identification of synovial markers of disease severity and poor response to therapy in early RA (Ref.22). In addition, using longitudinal synovial biopsy samples collected prospectively in patients prior to, and 3 months after initiation of therapy, we were able to identify synovial molecular targets of several therapies in RA : methotrexate, tocilizumab, adalimumab and also rituximab (Ref.23-26).While TNF blockade decreases expression of genes involved in cell proliferation in RA synovitis, the other drugs induce very similar molecular changes in the RA synovium, characterized by a decrease in IL6-dependent T cell activation (Ref.26).

   In the present project, we want to compare global molecular profiles up-or down-regulated in synovitis of patients with psoriatic arthritis, before and after targeted therapy. This project takes advantage of our strong experience in the field of molecular profiling of synovial biopsies, and evaluation of responses to biological agents (Ref.20-26).
2. STUDY QUESTION AND OBJECTIVES 2.1 STUDY QUESTION We intend to evaluate the global transcriptomic effects of Apremilast (Otezla®) in synovial biopsies from DMARD-naïve and biological-naive patients with psoriatic arthritis, obtained prior to and 24 weeks after initiation of therapy.

Identification of the synovial effects of Apremilast therapy in psoriatic arthritis will be a step forward in understanding not only the mode of action of the drug at the site of inflammation, but also in the identification of molecular patterns associated with good response to therapy. The main advantage of our approach compared to other biomarker studies, is that we use synovial material as such, and not peripheral blood, which is a more remote location in terms of cellular targets of the drug.

2.2 STUDY OBJECTIVES

Primary Objective To evaluate the global transcriptomic effects of apremilast in synovial biopsies of DMARD (cs and b) naïve PsA patients, obtained prior to, and 24 weeks after apremilast therapy.

Secondary Objective To correlate the molecular effects of apremilast therapy to clinical and ultrasound response, with a specific attention on joints, enthesis.

Evaluate clinical response at W24, by using ACR20/50/70 response criteria.

Identify candidate synovial markers/pathways associated with response to apremilast in PsA by correlating molecular signals at baseline with the clinical response observed at week 24.

2.3 STUDY DURATION The study duration is 36 months. Screening phase: up to 4 weeks Active treatment: 24 weeks Follow-up period: 4 weeks

* Screening period will start: October 2020
* Estimated first patient inclusion (FPI): November 2020
* Estimated last patient inclusion (LPI): January 2022
* Estimated last patient last visit (LPLV): december 2022
* Publication summary: dec 2023
* Final report: feb 2024

ELIGIBILITY:
Inclusion Criteria:

Patients who meet ALL the following criteria can be enrolled:

* Patient must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study assessment is performed.
* Male or non-pregnant, non-nursing female patients at least 18 years of age.
* With a diagnosis of active PsA according to CASPAR criteria
* Naïve to csDMARD and bDMARD,
* At least 1 swollen joint at screening or baseline (despite NSAIDs therapy) with ability to perform a synovial biopsy at W0.
* Concomitant oral steroids (no more than 10 mg/day of prednisolone), NSAIDs, or painkillers is permitted if started prior to the study and remain at a stable dose at least 4 weeks before the baseline.
* Allowed concomitant medications are to remain stable through week 24.
* At least one joint (small or large) to biopsy in order to get synovial tissue. Small joints must have an US scoring > 2 on grey-scale score/power Doppler.

Exclusion Criteria:

Patients who meet AT LEAST one of the following exclusion criteria will be excluded:

* Contraindications for needle-arthroscopy.
* Patients with hypersensitivity to apremilast or to one of its excipients
* Prior csDMARD or bDMARD therapy,
* Women who are pregnant, breastfeeding or planning on becoming pregnant for the 24 weeks of the drug administration,
* Non-menopausal women who are not using an adequate contraception method,
* Patients with conditions/concomitant diseases making them non evaluable for the primary endpoint
* Impossibility to meet specific protocol requirements (e.g. blood sampling)
* Patient is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Uncooperative or any condition that could make the patient potentially noncompliant to the study procedures
* Any therapy by intra-articular injections (e.g. corticosteroid) within 4 weeks before baseline.
* Any intramuscular corticosteroid injection within 4 weeks before baseline.
* A history of active tuberculosis (TB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Quantitative measurement of the molecular changes in relation to the up-regulated or down-regulated genes in the synovium. | 24 weeks
  The primary endpoint of the study is not the efficacy of the drug, but the molecular changes it induce in the synovium.
  In a first set of analyses, the magnitude of fold-changes in global gene expression profiles between baseline and W24 will be analysed. The higher values correspond to the high intensity in the up-regulation or down-regulation of the gene expression.

SECONDARY OUTCOMES:
Comparison between the magnitude of molecular changes (up-regulation or down-regulation of the genes) and clinical changes (improvement or worsening of the swollen joints count). | 24 weeks
  The swollen joints count (0 to 66) will be assessed. Lowered scores correspond to an improvement (remission or low disease activity), and increased value to a worsening of the clinical conditions (high disease activity). The value of the joints count will be compared to the magnitude of the up-regulation or down-regulation in the gene expression profiles.
Comparison between the magnitude of molecular changes (up-regulation or down-regulation of the genes) and imaging changes on Grey Scale ultrasound (GSUS). | 24 weeks
  Synovitis (inflammation in the synovium) is scored by US in Grey-Scale (GS) (0 to 3). 0 correspond to lack of inflammation, and 3 to high amount of inflammation. The US changes in GS will be compared to the magnitude of up-regulation or down-regulation in the gene expression profiles.
Comparison between the magnitude of molecular changes (up-regulation or down-regulation of the genes) and imaging changes on Power Doppler ultrasound (PDUS). | 24 weeks
  Synovitis (inflammation in the synovium) is scored by US with the Power Doppler (PD) (0 to 3). 0 correspond to lack of inflammation, and 3 to high amount of inflammation. The US changes in PD will be compared to the magnitude of up-regulation or down-regulation in the gene expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Adrien NZEUSSEU TOUKAP, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Adrien NZEUSSEU TOUKAP, Brussels, Belgium

REFERENCES:
- [Background] Ferrandiz C, Bordas X, Garcia-Patos V, Puig S, Pujol R, Smandia A. Prevalence of psoriasis in Spain (Epiderma Project: phase I). J Eur Acad Dermatol Venereol. 2001 Jan;15(1):20-3. doi: 10.1046/j.1468-3083.2001.00191.x. PMID 11451315
- [Background] Augustin M, Reich K, Glaeske G, Schaefer I, Radtke M. Co-morbidity and age-related prevalence of psoriasis: Analysis of health insurance data in Germany. Acta Derm Venereol. 2010 Mar;90(2):147-51. doi: 10.2340/00015555-0770. PMID 20169297
- [Background] Rodgers M, Epstein D, Bojke L, Yang H, Craig D, Fonseca T, Myers L, Bruce I, Chalmers R, Bujkiewicz S, Lai M, Cooper N, Abrams K, Spiegelhalter D, Sutton A, Sculpher M, Woolacott N. Etanercept, infliximab and adalimumab for the treatment of psoriatic arthritis: a systematic review and economic evaluation. Health Technol Assess. 2011 Feb;15(10):i-xxi, 1-329. doi: 10.3310/hta15100. PMID 21333232
- [Background] Moll JM, Wright V. Psoriatic arthritis. Semin Arthritis Rheum. 1973;3(1):55-78. doi: 10.1016/0049-0172(73)90035-8. No abstract available. PMID 4581554
- [Background] Kavanaugh A, Mease PJ, Gomez-Reino JJ, Adebajo AO, Wollenhaupt J, Gladman DD, Lespessailles E, Hall S, Hochfeld M, Hu C, Hough D, Stevens RM, Schett G. Treatment of psoriatic arthritis in a phase 3 randomised, placebo-controlled trial with apremilast, an oral phosphodiesterase 4 inhibitor. Ann Rheum Dis. 2014 Jun;73(6):1020-6. doi: 10.1136/annrheumdis-2013-205056. Epub 2014 Mar 4. PMID 24595547
- [Background] Wong K, Gladman DD, Husted J, Long JA, Farewell VT. Mortality studies in psoriatic arthritis: results from a single outpatient clinic. I. Causes and risk of death. Arthritis Rheum. 1997 Oct;40(10):1868-72. doi: 10.1002/art.1780401021. PMID 9336423
- [Background] Menter A, Korman NJ, Elmets CA, Feldman SR, Gelfand JM, Gordon KB, Gottlieb AB, Koo JY, Lebwohl M, Lim HW, Van Voorhees AS, Beutner KR, Bhushan R. Guidelines of care for the management of psoriasis and psoriatic arthritis: section 4. Guidelines of care for the management and treatment of psoriasis with traditional systemic agents. J Am Acad Dermatol. 2009 Sep;61(3):451-85. doi: 10.1016/j.jaad.2009.03.027. Epub 2009 Jun 3. PMID 19493586
- [Background] Schett G, Sloan VS, Stevens RM, Schafer P. Apremilast: a novel PDE4 inhibitor in the treatment of autoimmune and inflammatory diseases. Ther Adv Musculoskelet Dis. 2010 Oct;2(5):271-8. doi: 10.1177/1759720X10381432. PMID 22870453
- [Background] Busa S, Kavanaugh A. Drug safety evaluation of apremilast for treating psoriatic arthritis. Expert Opin Drug Saf. 2015 Jun;14(6):979-85. doi: 10.1517/14740338.2015.1031743. Epub 2015 Mar 31. PMID 25827658
- [Background] Schafer P. Apremilast mechanism of action and application to psoriasis and psoriatic arthritis. Biochem Pharmacol. 2012 Jun 15;83(12):1583-90. doi: 10.1016/j.bcp.2012.01.001. Epub 2012 Jan 10. PMID 22257911
- [Background] Gooderham M, Papp K. Selective Phosphodiesterase Inhibitors for Psoriasis: Focus on Apremilast. BioDrugs. 2015 Oct;29(5):327-39. doi: 10.1007/s40259-015-0144-3. PMID 26481941
- [Background] Schafer PH, Truzzi F, Parton A, Wu L, Kosek J, Zhang LH, Horan G, Saltari A, Quadri M, Lotti R, Marconi A, Pincelli C. Phosphodiesterase 4 in inflammatory diseases: Effects of apremilast in psoriatic blood and in dermal myofibroblasts through the PDE4/CD271 complex. Cell Signal. 2016 Jul;28(7):753-63. doi: 10.1016/j.cellsig.2016.01.007. Epub 2016 Jan 22. PMID 26806620
- [Background] Edwards CJ, Blanco FJ, Crowley J, Birbara CA, Jaworski J, Aelion J, Stevens RM, Vessey A, Zhan X, Bird P. Apremilast, an oral phosphodiesterase 4 inhibitor, in patients with psoriatic arthritis and current skin involvement: a phase III, randomised, controlled trial (PALACE 3). Ann Rheum Dis. 2016 Jun;75(6):1065-73. doi: 10.1136/annrheumdis-2015-207963. Epub 2016 Jan 20. PMID 26792812
- [Background] Papp K, Reich K, Leonardi CL, Kircik L, Chimenti S, Langley RG, Hu C, Stevens RM, Day RM, Gordon KB, Korman NJ, Griffiths CE. Apremilast, an oral phosphodiesterase 4 (PDE4) inhibitor, in patients with moderate to severe plaque psoriasis: Results of a phase III, randomized, controlled trial (Efficacy and Safety Trial Evaluating the Effects of Apremilast in Psoriasis [ESTEEM] 1). J Am Acad Dermatol. 2015 Jul;73(1):37-49. doi: 10.1016/j.jaad.2015.03.049. PMID 26089047
- [Background] Paul C, Cather J, Gooderham M, Poulin Y, Mrowietz U, Ferrandiz C, Crowley J, Hu C, Stevens RM, Shah K, Day RM, Girolomoni G, Gottlieb AB. Efficacy and safety of apremilast, an oral phosphodiesterase 4 inhibitor, in patients with moderate-to-severe plaque psoriasis over 52 weeks: a phase III, randomized controlled trial (ESTEEM 2). Br J Dermatol. 2015 Dec;173(6):1387-99. doi: 10.1111/bjd.14164. Epub 2015 Nov 7. PMID 26357944
- [Background] Ritchlin CT, Colbert RA, Gladman DD. Psoriatic Arthritis. N Engl J Med. 2017 Mar 9;376(10):957-970. doi: 10.1056/NEJMra1505557. No abstract available. PMID 28273019
- [Background] Nzeusseu Toukap A, Galant C, Theate I, Maudoux AL, Lories RJ, Houssiau FA, Lauwerys BR. Identification of distinct gene expression profiles in the synovium of patients with systemic lupus erythematosus. Arthritis Rheum. 2007 May;56(5):1579-88. doi: 10.1002/art.22578. PMID 17469140
- [Background] Lauwerys BR, Hernandez-Lobato D, Gramme P, Ducreux J, Dessy A, Focant I, Ambroise J, Bearzatto B, Nzeusseu Toukap A, Van den Eynde BJ, Elewaut D, Gala JL, Durez P, Houssiau FA, Helleputte T, Dupont P. Heterogeneity of synovial molecular patterns in patients with arthritis. PLoS One. 2015 Apr 30;10(4):e0122104. doi: 10.1371/journal.pone.0122104. eCollection 2015. PMID 25927832
- [Background] De Groof A, Ducreux J, Humby F, Nzeusseu Toukap A, Badot V, Pitzalis C, Houssiau FA, Durez P, Lauwerys BR. Higher expression of TNFalpha-induced genes in the synovium of patients with early rheumatoid arthritis correlates with disease activity, and predicts absence of response to first line therapy. Arthritis Res Ther. 2016 Jan 20;18:19. doi: 10.1186/s13075-016-0919-z. PMID 26792343
- [Background] Badot V, Galant C, Nzeusseu Toukap A, Theate I, Maudoux AL, Van den Eynde BJ, Durez P, Houssiau FA, Lauwerys BR. Gene expression profiling in the synovium identifies a predictive signature of absence of response to adalimumab therapy in rheumatoid arthritis. Arthritis Res Ther. 2009;11(2):R57. doi: 10.1186/ar2678. Epub 2009 Apr 23. PMID 19389237
- [Background] Badot V, Durez P, Van den Eynde BJ, Nzeusseu-Toukap A, Houssiau FA, Lauwerys BR. Rheumatoid arthritis synovial fibroblasts produce a soluble form of the interleukin-7 receptor in response to pro-inflammatory cytokines. J Cell Mol Med. 2011 Nov;15(11):2335-42. doi: 10.1111/j.1582-4934.2010.01228.x. PMID 21129157
- [Background] Gutierrez-Roelens I, Galant C, Theate I, Lories RJ, Durez P, Nzeusseu-Toukap A, Van den Eynde B, Houssiau FA, Lauwerys BR. Rituximab treatment induces the expression of genes involved in healing processes in the rheumatoid arthritis synovium. Arthritis Rheum. 2011 May;63(5):1246-54. doi: 10.1002/art.30292. PMID 21337318
- [Background] Ducreux J, Durez P, Galant C, Nzeusseu Toukap A, Van den Eynde B, Houssiau FA, Lauwerys BR. Global molecular effects of tocilizumab therapy in rheumatoid arthritis synovium. Arthritis Rheumatol. 2014 Jan;66(1):15-23. doi: 10.1002/art.38202. PMID 24449571
- See also: Federal Agency for Medicines and Health Products (famhp/afmps/fagg). Otezla (apremilast): nouvelles recommandations importantes concernant les idées et comportements suicidaires. — https://www.fagg-afmps.be/sites/default/files/dhpc_otezla_fr_-_website.pdf
- See also: Otezla (apremilast): Nieuw belangrijk advies met betrekking tot suïcidale ideatie en suïcidaal gedrag (28 oktober 2016). — https://www.fagg-afmps.be/sites/default/files/dhpc_otezla_nl_-_website.pdf